CLINICAL TRIAL: NCT01421589
Title: The Effects of Short Term Growth Hormone Treatment on Skeletal Muscle Phosphocreatine Recovery in Obesity
Brief Title: Growth Hormone Treatment on Phosphocreatine Recovery in Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Hideo Makimura, Principal Investigator, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011-P-000770
Record Dates: First submitted 2011-08-19; First posted 2011-08-23 (Estimated); Results first posted 2014-07-01 (Estimated); Last update posted 2014-07-01 (Estimated); Status verified 2014-05

CONDITIONS: Obese; Growth Hormone Secretion Abnormality
Keywords: Growth hormone; GH; Obesity; Mitochondrial function; reduced growth hormone secretion
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Growth Hormone (Experimental)
  Interventions: Drug: Growth hormone treatment

INTERVENTIONS:
Drug: Growth hormone treatment — Growth hormone 0.4 mg once daily (titrated to IGF-1) by sub-cutaneous injection for 12 weeks.

SUMMARY:
Obesity is associated with reduced growth hormone (GH) secretion. Reduced GH secretion in obesity is associated with increased cardiovascular disease risk. However, it is not yet known how reduced GH increases cardiovascular disease risk in obesity. The investigators hypothesize that reduced GH contributes to dysfunction of the mitochondria. Therefore, the investigators hypothesize that treatment of obese subjects with reduced GH secretion with GH will improve mitochondrial function and that this improvement in mitochondrial function will contribute, in part, to the effects of GH to improve metabolic parameters in obesity. The investigators propose to study skeletal muscle mitochondria in obese subjects with reduced GH secretion using magnetic resonance spectroscopy and muscle biopsies before and after treatment with GH.

ELIGIBILITY:
Inclusion Criteria:

1. Men age 18-60 years old
2. BMI ≥ 30 kg/m2
3. Waist circumference ≥ 102 cm
4. Peak GH value of ≤ 4.2 μg/l on standard GHRH-arginine stimulation test

Exclusion Criteria:

1. Obesity due to a known secondary cause (Cushing's syndrome, hypothyroidism, etc) or a history of gastric bypass procedure.
2. Subjects who have a known history of diabetes, fasting blood sugar >125 mg/dl or using any anti-diabetic drugs.
3. Use of Aspirin, Clopidogrel (Plavix), Warfarin (Coumadin) or other anti-coagulants
4. Subjects on testosterone, glucocorticoids, anabolic steroids, GHRH, GH or IGF-1 within 3 months of enrollment.
5. Changes in lipid lowering or anti-hypertensive regimen within 3 months of screening
6. History of pituitary tumor, hypopituitarism, pituitary surgery, pituitary/brain radiation or traumatic brain injury or any other condition known to affect the GH axis.
7. Severe chronic illness including HIV, active malignancy or history of colon cancer.
8. Hemoglobin < 9.0 g/dL, SGOT > 2.5 x upper limit normal, Creatinine >1.5 mg/dL, or PSA >5 ng/ml.
9. Subject is currently enrolled in another investigational device or drug trial(s), or subject has received other investigational agent(s) within 28 days of baseline visit.
10. Any condition judged by the patient's physician to cause this clinical trial to be detrimental to the patient.
11. Contraindications to MRI scanning.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2011-09; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hideo Makimura, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Growth Hormone Treatment: Growth hormone treatment: recombinant human Growth hormone 0.4 mg once daily (titrated to IGF-1) by sub-cutaneous injection for 12 weeks.
Period: Overall Study
Arm/Group | Growth Hormone Treatment
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Obese male subjects with reduced growth hormone secretion
Arm/Group | Growth Hormone
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.9 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 10
  More than one race | 0
  Unknown or Not Reported | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Phosphocreatine Recovery
Description: The primary objective of this study is to determine the effects of growth hormone on mitochondrial function as assessed by 31P-MRS in obese subjects with reduced GH secretion. Mitochondrial function was represented by ViPCr, a measure of phosphocreatine recovery after sub-maximal exercise. Univariate regression analyses was performed to assess the relationship between the change in skeletal muscle IGF-1 mRNA after 12 weeks treatment with rhGH to change in ViPCr.
Time Frame: 12-weeks
Population: All 15 subjects underwent 31P-MRS, however, two scans were not evaluable due to technical difficulties. In addition, paired analyses (both Baseline and 12-weeks) from only 10 subjects were available for gene expression analyses. Therefore univariate regression analyses between IGF-1 mRNA and PCr recovery could only be performed in 10 subjects.
Measure: Number; unit: correlation coefficient
Arm/Group | Growth Hormone Treatment
Number analyzed (Participants) | 10
correlation coefficient | 0.74 (5.4)
Statistical Analysis 1: Comparison: Growth Hormone Treatment; Univariate regression analyses was performed to assess the relationship between change in skeletal muscle IGF-1 mRNA expression after 12 weeks treatment with rhGH and change in ViPCr; Test type: Superiority or Other; p = 0.02, Regression, Linear

2. Secondary Outcome: Change in Circulating IGF-1 Concentration
Description: Change in circulating IGF-1 from Baseline to 12-weeks is reported.
Time Frame: Baseline and 12-weeks
Measure: Mean (Standard Error); unit: ug/l
Arm/Group | Growth Hormone Treatment
Number analyzed (Participants) | 15
ug/l | 218 (29)
Statistical Analysis 1: Comparison: Growth Hormone Treatment; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

3. Secondary Outcome: Change in Skeletal Muscle IGF-1 Gene Expression
Description: Change in skeletal muscle IGF-1 gene mRNA expression from Baseline to 12-weeks is reported.
Time Frame: Baseline and 12-weeks
Population: Paired analyses (both Baseline and 12-weeks) from only 10 subjects are available for gene expression
Measure: Mean (Standard Error); unit: fold change
Arm/Group | Growth Hormone Treatment
Number analyzed (Participants) | 10
fold change | 2.1 (0.3)
Statistical Analysis 1: Comparison: Growth Hormone Treatment; Test type: Superiority or Other; p < 0.05, t-test, 2 sided

4. Secondary Outcome: Change in Body Composition
Description: Change in waist circumference from Baseline to 12-weeks is reported.
Time Frame: Baseline and 12-weeks
Measure: Mean (Standard Error); unit: cm
Arm/Group | Growth Hormone Treatment
Number analyzed (Participants) | 15
cm | -3 (1)
Statistical Analysis 1: Comparison: Growth Hormone Treatment; Test type: Superiority or Other; p < 0.05, t-test, 2 sided

5. Secondary Outcome: Change in Inflammatory Marker
Description: Change in high sensitivity C-reactive protein (hsCRP) from Baseline to 12-weeks is reported.
Time Frame: Baseline and 12-weeks
Measure: Mean (Standard Error); unit: mg/l
Arm/Group | Growth Hormone Treatment
Number analyzed (Participants) | 15
mg/l | -1.78 (0.57)
Statistical Analysis 1: Comparison: Growth Hormone Treatment; Test type: Superiority or Other; p < 0.05, t-test, 2 sided

6. Secondary Outcome: Change in Insulin Sensitivity
Description: Change in fasting glucose from Baseline to 12-weeks is reported.
Time Frame: Baseline and 12-weeks
Measure: Mean (Standard Error); unit: mg/dl
Arm/Group | Growth Hormone Treatment
Number analyzed (Participants) | 15
mg/dl | 6 (3)
Statistical Analysis 1: Comparison: Growth Hormone Treatment; Test type: Superiority or Other; p < 0.05, t-test, 2 sided

7. Secondary Outcome: Change in Phosphocreatine Recovery
Description: Change in phosphocreatine recovery, represented by ViPCr, from Baseline to 12-weeks is reported.
Time Frame: Baseline and 12-weeks
Population: Obese men with reduced GH secretion were treated with rhGH for 12 weeks. All 15 subjects underwent 31P-MRS, however, two scans were not evaluable due to technical difficulties.
Measure: Mean (Standard Error); unit: mM/min
Groups:
- Growth Hormone: Growth hormone treatment: recombinant human Growth hormone 0.4 mg once daily (titrated to IGF-1) by sub-cutaneous injection for 12 weeks.
Arm/Group | Growth Hormone
Number analyzed (Participants) | 13
mM/min | -10.2 (7.5)
Statistical Analysis 1: Comparison: Growth Hormone; Test type: Superiority or Other; p > 0.05, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Growth Hormone Treatment
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 11/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Growth Hormone Treatment (N=15)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4
Carpal tunnel syndrome (Musculoskeletal and connective tissue disorders) | 0
Head ache (Nervous system disorders) | 2
Hypersensitivity reaction (Immune system disorders) | 0
Injection site bleeding (Skin and subcutaneous tissue disorders) | 1
Injection site bruising (Skin and subcutaneous tissue disorders) | 5
Injection site pain, pruritis, erythema, induration (Skin and subcutaneous tissue disorders) | 0
Myalgias (Musculoskeletal and connective tissue disorders) | 5
Paresthesias (Nervous system disorders) | 1
Peripheral edema (Cardiac disorders) | 4
Diabetes (Metabolism and nutrition disorders) | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less